CLINICAL TRIAL: NCT01491906
Title: Weight Loss Among Adults in Beijing, China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: The George Institute for Global Health, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A0458
Record Dates: First submitted 2011-12-06; First posted 2011-12-14 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Obesity; Hypertension
MeSH Terms: conditions — Obesity; Hypertension | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Text-Messaging (Experimental): The group that receives the behavioral counseling and text messaging lifestyle intervention
  Interventions: Behavioral: Text Messaging and Behavior Counseling
- Usual Care (No Intervention): This group will receive usual care

INTERVENTIONS:
Behavioral: Text Messaging and Behavior Counseling — Participants randomized to the intervention arm will receive a series of components, delivered over 6 months: personalized behavior change goals to be self-monitored via text messaging, group "starter" counseling sessions, and personalized individual counseling. Each participant will also receive a pedometer to facilitate self-monitoring.
  Arms: Text-Messaging

SUMMARY:
The purpose of this study is to test the effect of a mobile phone-assisted lifestyle intervention on weight loss at 6 months among overweight/obese Chinese adults, as compared to a control group.

DETAILED DESCRIPTION:
The rapid gains in China's economic development during the past two decades have been accompanied by similar gains in the population's waistline. Over 25% of Chinese adult females and more than a third of males are overweight or obese and rates are highest in urban areas such as Beijing. By 2015, overweight/obesity prevalence in China may reach 50% , thus imposing a heavy toll on chronic disease rates and health care costs. Despite these pressing public health challenges, very few obesity intervention studies have been conducted among Chinese adults.

Duke University and Peking University have partnered to implement an intervention to address these rapid changes in weight. 124 participants in Beijing will be randomly assigned to either: (1) usual care (UC), or; (2) a 6-month weight loss (WL) intervention condition. The primary outcome is weight change (kg) at 6 months post-baseline. Secondary outcomes include change in blood pressure, weight circumference, dietary intake, physical activity, and psychosocial mediators at 6 months post-baseline.

Participants randomized to the intervention arm will receive a series of components, delivered over 6 months: personalized behavior change goals to be self-monitored via text messaging, group "starter" counseling sessions, and personalized individual counseling. Each participant will also receive a pedometer to facilitate self-monitoring. These are evidence-based approaches, drawn from the investigators' collective research experience.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 24,
* age 30-55 years
* current use of a mobile phone
* interest in losing weight.

Exclusion Criteria:

* Pregnancy or plans to become pregnant within 10 months of recruitment
* current lactation
* occurrence of a major cardiovascular disease (e.g., myocardial infarction or stroke in the past 6 months)
* other serious medical conditions that contraindicate weight loss (e.g., end-stage renal disease on dialysis, cancer diagnosis or treatment in past 2 years)
* blood pressure ≥ 160/100 mm Hg
* type 2 diabetes or controlled by lifestyle only
* use of medications known to increase body weight
* substance abuse; psychiatric illness, including major depression, which could interfere with study adherence
* prior or planned bariatric surgery
* use of weight loss medications or weight loss ≥ 5% of initial weight in past 6 months
* plans to relocate in next 10 months

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 123 (Actual)
Dates: Start 2011-05; Primary Completion 2012-02 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Weight in kg | baseline and 6-months
  Weight measurements will be taken at baseline and at the 6-month follow-up visit

SECONDARY OUTCOMES:
Change in body composition & behavior | baseline and 6-months
  Secondary outcomes include change in blood pressure, weight circumference, dietary intake, physical activity, and psychosocial mediators at 6 months post-baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University, Beijing, China

REFERENCES:
- [Result] Lin PH, Wang Y, Levine E, Askew S, Lin S, Chang C, Sun J, Foley P, Wang H, Li X, Bennett GG. A text messaging-assisted randomized lifestyle weight loss clinical trial among overweight adults in Beijing. Obesity (Silver Spring). 2014 May;22(5):E29-37. doi: 10.1002/oby.20686. Epub 2014 Jan 9. PMID 24375969